CLINICAL TRIAL: NCT06942494
Title: Effect of a Family-Based Cognitive Behavioral Therapy Self-Help Intervention for Adolescents With Obsessive-Compulsive Disorder：A Randomized Controlled Trial
Brief Title: Effect of a Family-Based CBT Self-Help Intervention for Adolescents With OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-112
Record Dates: First submitted 2025-04-07; First posted 2025-04-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: Obsessive - Compulsive Disorder; Adolescents; Bibliotherapy
MeSH Terms: conditions — Compulsive Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-Based Self-Help Intervention Group (Experimental): Adolescents with OCD in this group will continue their stable pharmacological treatment for at least six weeks prior to enrollment. After baseline assessment, they will receive a 12-week structured cognitive behavioral therapy (CBT)-based self-help intervention, specifically designed for chinese adolescents and involving family participation. After the 12-week intervention, participants will enter a 3-month follow-up phase, during which no new therapeutic components will be introduced, but data on symptom maintenance and treatment adherence will be collected.During the 12-week intervention they will continue with the medications they already have.
  Interventions: Behavioral: Family-Based Self-help Book for Adolescents with Obsessive-Compulsive Disorder
- Treatment-As-Usual Waitlist Control Group (Active Comparator): Adolescents with OCD in this group will be similarly required to receive at least six weeks of stabilizing medication prior to enrollment. In this group, participants will be treated as usual. Namely, they will continue with the medications they already have with no changes throughout the 12-week intervention period. No psychological intervention will be provided during this phase. After completing the follow-up assessment at week 12, participants will be offered access to the CBT-based self-help book as a delayed intervention.
  Interventions: Drug: conventional medical treatment (TAU)

INTERVENTIONS:
Drug: conventional medical treatment (TAU) — In this study, the investigators use selective serotonin reuptake inhibitors (SSRIs, i.e., sertraline, fluoxetine and fluvoxamine)and tricyclic drugs(i.e., clomipramine) approved by the State Food and Drug Administration (CFDA) for the treatment of OCD in children and adolescents. The drugs used in this study are commonly used in clinical practice and have a good safety profile. The maximum dosage shall not exceed the maximum dosage prescribed in the instruction manual, or the maximum dosage tolerated by the patients.
  Arms: Treatment-As-Usual Waitlist Control Group
Behavioral: Family-Based Self-help Book for Adolescents with Obsessive-Compulsive Disorder — The self-help book used in this study was independently developed by members of our research team. Its content is based on Exposure and Response Prevention (ERP). Adolescent patients with OCD will be instructed to read one chapter of the self-help book each week and complete the corresponding exercises. This 12-week intervention will involve self-guided practice conducted by the adolescent and their family members.Throughout the intervention period, adolescents and their caregivers may contact the therapist via WeChat to ask questions and upload records of their completed exercises. The therapist will respond to any questions within 48 hours by sending written messages via WeChat, with each family receiving no more than 30 minutes of such written guidance per week. All therapists will be required to keep a weekly log of the time spent providing guidance to each participating family.If a participating family does not initiate contact, the therapist will not provide proactive guidance.
  Arms: Family-Based Self-Help Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if self-help book can be used to treat obsessive-compulsive disorder (OCD) in adolescents aged 10 to 17. The main questions it aims to answer are:

Can adolescents and their parents effectively reduce the severity of the obsessive-compulsive symptoms in adolescents who are already stably taking medications through self-help books? What are the characteristics of adolescents who are best suited to use self-help intervention book to treat obsessive-compulsive symptoms?

Researchers will compare the use of a self-help books plus medication with medication alone to see if the combination of the self-help intervention and drug treatment can improve the obsessive-compulsive symptoms of adolescents more effectively.

Participants will:

* Read one chapter of a self-help book and complete the corresponding exercise each week for 12 weeks
* Visit the clinic before and after intervention for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 17 years
2. Satisfied with the diagnostic criteria for OCD in DSM-5
3. 16≤CY-BOCS score ≤23
4. Taking medication stably for 6 weeks
5. Education level ⩾6 years
6. At least one parent can accompany the patients throughout the entire intervention process
7. The patient and the participating parent have sufficient reading and writing skills to complete the treatment intervention
8. The patient and the participating parent have adequate auditory and visual abilities skills to complete the necessary examinations for the study

(7) Right-handed (this criterion is for fMRI subjects only) (8) Subjects and their guardians understood the study and signed informed consent.

Exclusion Criteria:

1. Obsessive-compulsive symptoms were too severe to participate in the experiment(CY-BOCS score ≥24)
2. High risk of suicide
3. Comorbid brain organic diseases, severe somatic diseases, learning disabilities, autism spectrum disorders, schizophrenia spectrum and other psychotic disorders, bipolar disorder, severe eating disorders, or substance abuse
4. Completed a Cognitive Behavioral Therapy (CBT) course for OCD within the past 12 months.
5. An IQ lower than 80
6. Currently undergoing other psychological/physical treatments
7. Uncooperative or unable to complete treatment
8. With metal implants in the body, such as pacemakers, intracranial silver clips, metal dentures, arterial stents, arterial clips, joint metal fixation, or other metal implants, etc. (this criterion is for fMRI subjects only)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The CY-BOCS is a clinician-rated instrument used to assess the severity of obsessive-compulsive symptoms in children and adolescents, which has good reliability and validity.. The total score ranges from 0 to 40, with higher scores indicating greater severity. The primary outcome is the change in CY-BOCS total score from baseline to each follow-up point.

SECONDARY OUTCOMES:
Change in Children's Depression Inventory (CDI) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The CDI is currently one of the most widely used self-assessment tools for evaluating depressive symptoms in children and adolescents. The scale consists of 27 multiple-choice items that assess a range of common depressive symptoms in youth, including sadness, hopelessness, suicidal ideation, and disturbances in sleep and appetite. Each item offers three response options reflecting increasing levels of symptom severity, scored as 0, 1, or 2.Scores range from 0 to 54, with higher scores indicating more severe depressive symptoms.The Chinese version used in the current study has demonstrated good psychometric properties, including a Cronbach's alpha of 0.85, a split-half reliability coefficient of 0.71, and a test-retest reliability coefficient of 0.75.
Change in Obsessive-Compulsive Inventory - Child Version (OCI-CV) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The Obsessive-Compulsive Inventory-Child Version (OCI-CV) is a multidimensional self-report scale developed by Foa and colleagues to assess the severity of obsessive-compulsive symptoms in children and adolescents aged 7 to 17. The scale consists of 21 items covering six symptom dimensions: Doubting/Checking, Obsessing, Hoarding, Washing, Ordering, and Neutralizing. Each item is rated on a 3-point Likert scale: 0 = Never, 1 = Sometimes, 2 = Always. The Chinese version of the scale used in current study has demonstrated strong psychometric properties and has been validated in international clinical samples. The internal consistency of the total scale was 0.856, and the internal consistency coefficients for the subscales ranged from 0.462 to 0.747. Test-retest reliability coefficients ranged from 0.532 to 0.758.The outcome is measured by the change in total score from baseline.
Change in Screen for Child Anxiety Related Emotional Disorders (SCARED) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The Screen for Child Anxiety Related Emotional Disorders (SCARED) is a self-report screening tool developed to assess anxiety symptoms in children and adolescents aged 9 to 18. It is widely used in clinical settings, research, and epidemiological studies as a supplemental tool for the diagnosis of anxiety-related disorders. The SCARED scale assesses five factors: somatization, generalized anxiety, separation anxiety, social phobia, and school phobia. Items are rated on a 3-point Likert scale: 0 = not true or hardly ever true, 1 = somewhat true or sometimes true, and 2 = very true or often true.
  The psychometric properties of the Chinese version used in the present study include test-retest reliability coefficients ranging from 0.567 to 0.608, split-half reliability of 0.88, and Cronbach's alpha coefficients ranging from 0.43 to 0.89. Item-total correlations ranged from 0.43 to 0.74.
Clinical Global Impression - Improvement (CGI-I) | Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The Clinical Global Impression (CGI) scale is a clinician-rated tool commonly used in psychiatric treatment studies to subjectively assess the severity of illness, treatment response, and overall therapeutic efficacy. It was developed by the Early Clinical Drug Evaluation Program (ECDEU) research group for clinical trials sponsored by the National Institute of Mental Health (NIMH). The CGI provides a clinician-based evaluation framework for determining the severity of a patient's symptoms and monitoring treatment progress over time. The CGI-I is used to assess overall improvement relative to baseline, scored from 1 (very much improved) to 7 (very much worse).
Clinical Global Impression - Severity (CGI-S) | Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The CGI-S is a clinician-rated measure of the severity of the patient's illness, scored from 1 (normal) to 7 (among the most extremely ill).

OTHER OUTCOMES:
Change in Family Accommodation Scale - Self-Rated Version (FAS-SR) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The Family Accommodation Scale-Self-Rated (FAS-SR) is a self-report instrument designed to assess the extent to which family members engage in accommodating behaviors related to a relative's obsessive-compulsive disorder (OCD).It comprises 19 items that measure various accommodating behaviors, such as providing reassurance, facilitating avoidance, and modifying routines to accommodate the OCD-affected individual. Each item is rated on a 5-point Likert scale, reflecting the frequency of the behavior over the past week. The scale has demonstrated excellent internal consistency, with a Cronbach's alpha of 0.91, and strong test-retest reliability (Intraclass Correlation Coefficient = 0.93) in clinical studies.The outcome is measured by the change in total score from baseline.
Change in Children's Obsessive-Compulsive Impact Scale - Revised (COIS-R) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The scale was developed to assess functional impairments specifically resulting from OCD. It consists of two versions: a child self-report and a parent-report, which differ only in pronoun usage ("you" for the child version; "your child" for the parent version).The instrument includes 33 items.Each item is rated on a 4-point Likert scale, where 0 indicates "no interference" and 3 indicates "severe interference." Higher total scores reflect greater functional impairment due to OCD symptoms. The original versions of both the parent and child reports demonstrated good internal consistency (Cronbach's alpha = 0.83-0.91 for the parent version; 0.78-0.92 for the child version) and test-retest reliability (Intraclass Correlation Coefficient = 0.81 for the parent version; 0.89 for the child version).The outcome is measured by the change in total score from baseline.
Change in Parenting Stress Index - Short Form (PSI-SF) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  The Parenting Stress Index-Short Form (PSI-SF) was developed to assess the level of parenting stress experienced by parents of children. The scale consists of three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, with each subscale comprising 12 items, for a total of 36 items.Items are rated on a 5-point Likert scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). The total score ranges from 36 to 180, with higher scores indicating greater parenting stress.Based on the total score, parenting stress is categorized into four levels: scores ≤85 indicate a normal range, 86-90 indicate a borderline level, 91-98 indicate a high level, and scores ≥99 reflect a very high level of stress. A total score above 90 suggests the need for psychological support from a mental health professional.The outcome is measured by the change in total score from baseline.
Change in Family Quality of Life Questionnaire (FAMQOL) Total Score | Baseline, Week 12 (post-intervention), Week 16 (1-month follow-up), Week 24 (3-month follow-up)
  This scale is designed to assess the quality of life of family caregivers. It consists of 16 items covering four dimensions: physical, social, spiritual, and psychological well-being. Each item is rated on a 5-point Likert scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Total scores range from 16 to 80, with higher scores indicating better quality of life among caregi is designed to assess the quality of life of family caregivers.The Chinese version used in the current study also showed good reliability and validity, with a Cronbach's α of 0.84.
Cost-effectiveness analysis | From Baseline to Week 12(post-treatment)
  The study designs a self-rated questionnaire about cost-effectiveness analyses, including both direct and indirect costs, and the caregivers of the patients fill out the questionnaire based on the bill. The cost-effectiveness analysis method (CEA) is used to measure the spending of three groups. The results of the total cost divided by CY-BOCS total reduction scores can reflect the cost required to obtain each unit of curative effect.
Dropout rate | From Baseline to Week 12(post-treatment)
  Dropout rate is recorded to evaluate treatment acceptability.
Homework completion | From Baseline to Week 12(post-treatment)
  Homework completion is recorded to evaluate treatment acceptability. The investigators use sign-in sheets to keep track of patients' homework completion.
Subjective satisfaction with treatment | From Baseline to Week 12(post-treatment)
  Subjective satisfaction with treatment is recorded to evaluate treatment acceptability. The investigators use a self-rated question（"Overall, how satisfied are you with your current treatment?") to measure patients' subjective satisfaction. The rating was done on a 7-item scale ranging from "Extremely dissatisfied" to "Extremely satisfied".
Treatment safety | From Baseline to Week 12(post-treatment)
  Adverse events (AEs) are the treatment safety indicators.
The University of Rhode Island Change Assessment(URICA) | Change from Baseline at Week12(post-treatment)
  The University of Rhode Island Change Assessment (URICA) is a self-report measurement method developed by McConnaughy, DiClemente, Prochaska, and Velicer . The 24-item version consists of four dimensions: Precontemplation (Cronbach's α = 0.79), Contemplation (Cronbach's α = 0.84), Action (Cronbach's α = 0.84), and Maintenance (Cronbach's α = 0.82). URICA is commonly used to study motivation related to the treatment of behavioral health issues, and few studies have explored the specific relationship between the URICA scales and Cognitive Behavioral Therapy (CBT) for obsessive-compulsive disorder.For the general population, the following cut-off scores may be appropriate: 8 or lower classified as People in Precontemplation 8-11 classified as People in Contemplation 11-14 classified as People in Preparation or Action For intensive service populations, it may be more appropriate to use only score in the range of 12-14 to classify those in preparation and action.
Short-Form 6-Dimension Health Survey Version 2 (SF-6Dv2) | From Baseline to Week 12(post-treatment)
  The full name of the self-completed Six-Dimension Health Survey Brief Form (SF-6Dv2) is "Short Form Six-Dimensions version 2". The SF-6Dv2 is an updated version of the widely used SF-36 Health Survey Questionnaire. It is a health utility measurement tool used to assess an individual's health-related quality of life (HRQoL) and convert it into health utility values, which can be used to calculate Quality Adjusted Life Years (QALYs). The SF-6Dv2 includes six dimensions: physical function, role limitation, social function, pain, mental health, and vitality.
Cost-utility analysis | From Baseline to Week 12(post-treatment)
  The cost-utility analysis method is used to measure the spending of improving patients' quality of life. The results of the total cost divided by SF-6Dv2 total improvement scores can reflect the cost required to obtain each unit of utility.
Change in Neuroelectrophysiological Indicators | Drug-free phase（before baseline and prior to starting medication）, Baseline at enrollment(Week 0), Post-Treatment(Week 12)
  The investigators will use the Go/No-Go and Flanker task as electroencephalography (EEG) task paradigms to assess the neuroelectrophysiological changes cauesd by self-help intervention in adolescents patients with OCD.
Change in Neuroimaging Indicators | Drug-free phase（before baseline and prior to starting medication）, Baseline at enrollment(Week 0), Post-Treatment(Week 12)
  The investigators will use structural and functional magnetic resonance imaging (MRI) to assess the neurophysiological changes cauesd by self-help intervention in adolescents patients with OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Doctor, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Xuhui, Shanghai Municipality, China